CLINICAL TRIAL: NCT05695014
Title: On the Effect of Discharge Education on Discharge Readiness and Satisfaction Given by Teach Back Method to Patients With Lumbar Disc Herniation Surgery
Brief Title: Effect of Discharge Education on Discharge Readiness and Satisfaction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Principal Investigator, Sevinç Taştan, Principal Investigator, Eastern Mediterranean University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: AG-1
Record Dates: First submitted 2023-01-13; First posted 2023-01-23 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Disc Herniation
Keywords: "discharge education"; "teach back metod"; "patients"
MeSH Terms: conditions — Intervertebral Disc Displacement

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Teach Back Metod (Experimental): The patients in the intervention group, on the other hand, will be trained with the teach-back method after completing the Personal Data Collection Form, Knowledge Test, and the "Ready to Discharge Scale". In these trainings, "Discharge Training Booklet", which will be prepared by the researcher, will be used as training material. This booklet will include information about discharge after Lumbar Disc Herniation Surgery.
  Interventions: Other: Teach Back Metod
- Control (No Intervention): The discharge training of the patients in the control group will be given by the health professionals responsible for their care and treatment according to their clinical routines.

INTERVENTIONS:
Other: Teach Back Metod — teach-back method is a way of checking understanding by asking patients to state in their own words what they need to know or do about their health. It is a way to confirm that you have explained things in a manner your patients understand.
  Arms: Teach Back Metod

SUMMARY:
Today, the increase in the cost of health services, the development of technology and the shortening of the hospitalization period day by day due to the reasons for preventing complications such as hospital infections have increased the importance of discharge planning. Optimum maintenance of home care of patients who underwent surgery after discharge is possible with an effective discharge education given to the patient and their relatives and the preparation of the patients. In this study, it was aimed to examine the effect of the discharge training given to the patients who underwent Lumbar Disc Herniation Surgery with the method of feedback on their readiness for discharge and their satisfaction with the discharge training.

Among the patient groups who were given and not trained by the teach-back method; H01. There is no difference between the scores of readiness for discharge. H02. There is no difference between discharge training satisfaction scores. H11: There is a difference between the scores of being ready for discharge. H12: There is a difference between discharge training satisfaction scores.

DETAILED DESCRIPTION:
While the discharge plan and education of the surgical patient constitute an important part of nursing care, it is also an indispensable element in improving the patient's quality of life. Early discharge training after lumbar disc herniation surgery relieves the patient's anxiety and facilitates compliance with the treatment. Patients' readiness for discharge includes adequate recovery for safe discharge, physical stability, functional ability, ability to manage self-care at home, and coping skills. The primary aim of this study is to examine the effect of discharge training given by the Teach Back Method on patients with lumbar disc herniation surgery on their readiness for discharge. The second aim of the study is to determine the satisfaction of the patients in the group using the Teach Back Method at discharge training.

Method Study design and setting: This randomized controlled trial will conduct at the Neurosurgery Service of Famagusta State Hospital and the Neurosurgery Clinic of the Nicosia Doctor Burhan Nalbantoglu State Hospital.

Sampling: The sample size of the study, the significance level of the hypothesis and the effect size were taken into account and the statistical power calculation related to the analyzes was made on the G Power 3.1.9.4 computer program. In the calculation made, the number of units in the sample was calculated as at least 68 people, 34 in each group, under the assump tions of 95% confidence interval, 80% power, and effect size 0.50.

Randomization: Allocation software was used to allocate the participants into two groups with equal numbers. Patients who meet the inclusion criteria of the study will be interviewed in the patient room by the researcher at the time of their admission to the hospital, and written and verbal consents will be obtained from the patients. Patients will then be included in the control or intervention group according to the randomization table.

Intervention: For the patients in the control group, the Personal Data Collection Form and the Readiness to Discharge Scale and Knowledge test will be filled. The discharge training of the patients in the control group will be given by the health professionals responsible for their care and treatment according to their clinical routines. The patients in the intervention group, on the other hand, will be trained with the teach-back method after completing the Personal Data Collection Form, Knowledge Test, and the "Ready to Discharge Scale". In these trainings, "Discharge Training Booklet", which will be prepared by the researcher, will be used as training material. This booklet will include information about discharge after Lumbar Disc Herniation Surgery. Expert opinion will be taken for the booklet. On the day of discharge, the patients in both groups will be given the 'Ready to Discharge Scale' and the 'Discharge Training Satisfaction Scale' and Knowledge Test.

Data Collection Tools The data collection tools to be used in the research consist of four parts. In the first part, "Descriptive information form" which includes information about patients and the disease, "Discharge Training Satisfaction Scale" in the second part, "Ready to Discharge Scale" in the third part lastly there is a knowledge test prepared to evaluate the effectiveness of the discharge training given in the fourth part.

Descriptive information form: This form of patients; It is a data collection tool that includes socio-demographic characteristics such as date of birth, gender, marital status, education level, and items related to the patient's disease.

Discharge Training Satisfaction Scale: The scale was developed by Meşe and Köşgeroğlu in 2021. It consists of 21 items. The Cronbach α reliability coefficient for the overall scale was found to be 0.91. The scale was designed as a 5-point Likert scale. The scores that can be obtained from the scale range from 21 to 105. The scale has no cut off.

Scale of Readiness to Discharge: The short form (Readiness for Hospital Discharge Scale/Short Form) developed by Weiss and et al. in 2014 was used. The scale consists of eight items and four dimensions, and items in the scale are evaluated on a scale ranging from 0 to 10, and higher scores indicate greater readiness.

Discharge training knowledge test: In line with the literature, a knowledge test consisting of 20-25 questions will be prepared for the content of the discharge training. In this knowledge test, there will be questions containing correct and incorrect answers, and patients will be expected to tick True, False and No idea. Expert opinion will be taken about the knowledge test.

Statistical analysis Collected data will analyse using the Statistical Package for Social Sciences (SPSS) version 24.0 (IBM, Armonk, NY, USA). Descriptive characteristics of the participants will be presented by the frequency of the responses. Descriptive statistics, including mean, standard deviation, and minimum and maximum values, will be used to present the scores obtained from the scales and the knowledge questionnaire. The Kolmogorov-Smirnov test will be used to examine the suitability of the data for normal distribution. Pearson's chi-squared test and Fisher's exact test will be used to compare descriptive characteristics. If it fits the normal distribution, parametric tests will be used. If it does not fit the normal distribution, nonparametric tests will be used.

ELIGIBILITY:
Inclusion Criteria:

over 18 years old Having undergone Lumbar Disc Herniation surgery, Patients who have the capacity to read and understand research guidelines

Exclusion Criteria:

Those who do not agree to participate in the research, Patients undergoing emergency surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2023-01-02 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
readiness for discharge | Change in Baseline readiness for discharge score at four days
  Readiness to Discharge Scale will be used examine the effect of discharge training given by the Teach Back Method on patients with lumbar disc herniation surgery on their readiness for discharge.

SECONDARY OUTCOMES:
Knowledge test | Change in Baseline Patient knowledge test at four days
  The discharge education knowledge test will be used to evaluate the patients' knowledge about their care in the post-discharge period.

CONTACTS AND LOCATIONS:
Overall Officials: Sevinc Tastan, Prof. Dr., Principal Investigator — Eastern Mediterranean University, Health Sciences Faculty
Locations (1):
- Eastern Mediterranean University, Health Sciences Faculty, Nursing Department, Famagusta, None Selected, Cyprus

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] He Q, Zhao J, Fan M, Wang F. Effect of continuous nursing based on wechat platform on postoperative rehabilitation of patients with lumbar disc herniation. Jpn J Nurs Sci. 2021 Apr;18(2):e12382. doi: 10.1111/jjns.12382. Epub 2020 Sep 28. PMID 32985089
- [Result] Moliterno JA, Knopman J, Parikh K, Cohan JN, Huang QD, Aaker GD, Grivoyannis AD, Patel AR, Hartl R, Boockvar JA. Results and risk factors for recurrence following single-level tubular lumbar microdiscectomy. J Neurosurg Spine. 2010 Jun;12(6):680-6. doi: 10.3171/2009.12.SPINE08843. PMID 20515355
- [Result] Talevski J, Wong Shee A, Rasmussen B, Kemp G, Beauchamp A. Teach-back: A systematic review of implementation and impacts. PLoS One. 2020 Apr 14;15(4):e0231350. doi: 10.1371/journal.pone.0231350. eCollection 2020. PMID 32287296
- [Result] Bahri N, Saljooghi S, Noghabi AD, Moshki M. Effectiveness of the teach-back method in improving self-care activities in postmenopausal women. Prz Menopauzalny. 2018 Mar;17(1):5-10. doi: 10.5114/pm.2018.74896. Epub 2018 Apr 11. PMID 29725278
- [Result] Shersher V, Haines TP, Sturgiss L, Weller C, Williams C. Definitions and use of the teach-back method in healthcare consultations with patients: A systematic review and thematic synthesis. Patient Educ Couns. 2021 Jan;104(1):118-129. doi: 10.1016/j.pec.2020.07.026. Epub 2020 Aug 1. PMID 32798080
- [Result] Prochnow JA, Meiers SJ, Scheckel MM. Improving Patient and Caregiver New Medication Education Using an Innovative Teach-back Toolkit. J Nurs Care Qual. 2019 Apr/Jun;34(2):101-106. doi: 10.1097/NCQ.0000000000000342. PMID 30198943
- [Result] Oh EG, Lee HJ, Yang YL, Kim YM. Effectiveness of Discharge Education With the Teach-Back Method on 30-Day Readmission: A Systematic Review. J Patient Saf. 2021 Jun 1;17(4):305-310. doi: 10.1097/PTS.0000000000000596. PMID 30882616
- [Result] Mollazadeh F MS, Hemmati Maslakpak M PhD. The Effect of Teach-Back Training on Self Management in Kidney Transplant Recipients: A Clinical Trial. Int J Community Based Nurs Midwifery. 2018 Apr;6(2):146-155. PMID 29607343
- [Result] Choi S, Choi J. Effects of the teach-back method among cancer patients: a systematic review of the literature. Support Care Cancer. 2021 Dec;29(12):7259-7268. doi: 10.1007/s00520-021-06445-w. Epub 2021 Jul 24. PMID 34302545
- [Result] Chandar JJ, Ludwig DA, Aguirre J, Mattiazzi A, Bielecka M, Defreitas M, Delamater AM. Assessing the link between modified 'Teach Back' method and improvement in knowledge of the medical regimen among youth with kidney transplants: The application of digital media. Patient Educ Couns. 2019 May;102(5):1035-1039. doi: 10.1016/j.pec.2018.12.007. Epub 2018 Dec 12. PMID 30622001
- [Result] Zabolypour S, Alishapour M, Behnammoghadam M, Abbasi Larki R, Zoladl M. A Comparison of the Effects of Teach-Back and Motivational Interviewing on the Adherence to Medical Regimen in Patients with Hypertension. Patient Prefer Adherence. 2020 Feb 26;14:401-410. doi: 10.2147/PPA.S231716. eCollection 2020. PMID 32161450
- [Result] Ghorbani B, Jackson AC, Noorchenarboo M, Mandegar MH, Sharifi F, Mirmoghtadaie Z, Bahramnezhad F. Comparing the Effects of Gamification and Teach-Back Training Methods on Adherence to a Therapeutic Regimen in Patients After Coronary Artery Bypass Graft Surgery: Randomized Clinical Trial. J Med Internet Res. 2021 Dec 10;23(12):e22557. doi: 10.2196/22557. PMID 34890346
- [Derived] Gullet A, Tastan S. The Effect of Discharge Training Based on Teach-Back Method on Discharge Readiness and Satisfaction: A Randomized Controlled Trial. Worldviews Evid Based Nurs. 2025 Aug;22(4):e70062. doi: 10.1111/wvn.70062. PMID 40698847